CLINICAL TRIAL: NCT01174563
Title: A Multi-Center Study Investigating the Correlation Between TARCEVA ®-Induced Rash and Efficacy Among EGFR-mutated NSCLC Patients Receiving First-line Therapy
Brief Title: A Study on the Correlation Between Tarceva (Erlotinib) - Induced Rash and Efficacy in EGFR Mutated Participants With Advanced Non-Small Cell Lung Cancer Receiving First-Line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25200
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg orally daily, with dose-reductions to 100 mg or 50 mg orally daily according to protocol

SUMMARY:
This open-label, single arm study will assess the correlation between Tarceva (erlotinib)-induced rash and efficacy in participants with inoperable, locally advanced, recurrent or metastatic non-small cell lung cancer (NSCLC) receiving first-line therapy for advanced disease. Participants will receive Tarceva at a dose of 150 mg daily orally, with dose adjustments according to protocol depending on toxicity. Anticipated time on study treatment is until disease progression, unacceptable toxicity, or withdrawal due to any reason.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Inoperable, locally advanced, recurrent or metastatic (Stage IIIB or IV) non-small cell lung cancer (NSCLC)
* Presence of epidermal growth factor receptor (EGFR) mutations
* Previously untreated with any systemic anti-neoplastic therapy for advanced disease
* Last dose of a prior systemic anti-neoplastic therapy for early-stage disease >/= 4 weeks before study start, and patient recovered from acute toxicities of any previous therapy
* A life expectancy of at least 12 weeks
* Able to comply with the study and its follow-up procedures
* Female participants had to be postmenopausal (24 months of amenorrhea), surgically sterile or agree to use a physical method of contraception. Male participants had to be surgically sterile or agree to use a barrier method of contraception. Women with an intact uterus (unless amenorrhoeic for the last 24 months) had to have a negative pregnancy test (urine or serum) within 3 days prior to erlotinib treatment initiation in the study. Male and female participants had to use effective contraception during the study and for a period of 90 days following the last administration of erlotinib. Acceptable methods of contraception included an established hormonal therapy or intrauterine device for females, and the use of a barrier contraceptive (i.e. diaphragm or condoms)

Exclusion Criteria:

* Pregnant or breast feeding women
* Granulocyte count <1.5 x 109/L and platelet count <100*10^9/L
* Serum bilirubin >1.5 upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2 * ULN (or >5 * ULN if clearly attributable to liver metastasis)
* Serum creatinine >1.5 ULN or creatinine clearance <60 mL/min
* Known allergy or other adverse reaction to study drug or any other related compound
* Any significant unstable systemic disease (including active infection, grade 4 hypertension, unstable angina, congestive heart failure, hepatic, renal or metabolic disease)
* Prior systemic anti-neoplastic therapy with HER1/EGFR inhibitors (as small molecule or monoclonal antibody therapy)
* Newly diagnosed or not yet definitively treated (i.e. stable disease >/= 2 months) CNS metastases or spinal cord compression
* Any significant ophthalmological abnormality, especially those likely to increase the risk of corneal epithelial lesions (the use of contact lenses is not recommended during the study)
* Participants who could not take oral medication, who required intravenous alimentation, had had prior surgical procedures affecting absorption, or had active peptic ulcer disease
* Active cancer other than NSCLC, except for basal cell or squamous cell carcinomas of the skin that have been excised and cured

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Israel (16):
  - Haemek Hospital; Oncology, Afula
  - Barzilai; Oncology, Ashkelon
  - Soroka Medical Center; Oncology Dept, Beersheba
  - Carmel Hospital; Oncology Unit, Haifa
  - Rambam Medical Center; Oncology, Haifa
  - Wolfson Hospital; Oncology, Holon
  - Shaare Zedek Medical Center; Oncology Dept, Jerusalem
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Nahariya Hospital; Oncology, Nahariya
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
  - Kaplan Medical Center; Oncology Inst., Rehovot
  - Ziv Medical Center; Oncology Department, Sefad
  - Sourasky / Ichilov Hospital; Oncology Department, Tel Aviv
  - Poria Hospital; Oncology, Tiberias
  - Assaf Harofeh; Oncology, Ẕerifin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 60 participants were enrolled in the study from 12 centers across Israel.
Groups:
- Erlotinib: Participants received 150 milligrams (mg) of Erlotinib orally daily, from Day 1 of the treatment period until unacceptable toxicity, disease progression or withdrawal due to any reason.
Period: Overall Study
Arm/Group | Erlotinib
Started | 60
Efficacy Set (Efficacy set included all participants who received at least one dose of study medication.) | 59
Safety Set (Safety set included all participants who received at least one dose of study medication.) | 59
Completed | 0
Not Completed | 60
Not completed — Progressive Disease | 45
Not completed — Death | 5
Not completed — Investigator's Discretion | 5
Not completed — Participant Withdrew Consent | 3
Not completed — Rash Adverse Event | 1
Not completed — Sponsor's decision | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Arm/Group | Erlotinib
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) According to Grade of Rash
Description: PFS was defined as the time from start of treatment to the date of the first documented progression according to revised Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 or the date of death for any reason in the absence of progressive disease (PD). Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: Day 1 of treatment period until disease progression or death (approximately up to 67 months)
Population: Efficacy set included all participants who received at least one dose of study drug. Here, "Number Analyzed" represents the number of participants who were evaluable at specified time points.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 59
months
  Grade 0: number analyzed (Participants) | 4
  Grade 0 | 2.16 [1.51 to NA] — Upper limit of 95% CI for Grade 0 was not estimated due to low number of participants with the events.
  Grade 1: number analyzed (Participants) | 13
  Grade 1 | 6.62 [3.57 to 13.48]
  Grade 2: number analyzed (Participants) | 23
  Grade 2 | 10.00 [7.31 to 23.61]
  Grade 3: number analyzed (Participants) | 19
  Grade 3 | 15.28 [10.62 to 25.77]
Statistical Analysis 1: Comparison: Erlotinib; Test type: Superiority; p = 0.005, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.41 to 0.83]

2. Secondary Outcome: Percentage of Participants With Erlotinib Dose Reductions Due to Rash Grade 3-4
Time Frame: Day 1 of treatment period until disease progression or death (approximately up to 67 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 59
percentage of participants
  Rash Grade III: number analyzed (Participants) | 19
  Rash Grade III | 8.5
  Rash Grade IV: number analyzed (Participants) | 0

3. Secondary Outcome: Progression-Free Survival (PFS) in Participants With Erlotinib Dose Reductions Due to Rash Grade 3-4
Description: as for outcome 1
Time Frame: Day 1 of treatment period until disease progression or death (approximately up to 67 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 59
months
  Rash grade III: number analyzed (Participants) | 19
  Rash grade III | 13.72 [7.31 to 50.13]
  Rash Grade IV: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent form up to end of study (approximately up to 67 months)
Description: An Adverse Event (AE) can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 4/59
Serious Adverse Events (participants affected / at risk) | 19/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=59)
Bradycardia (Cardiac disorders) | 1
Vision blurred (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroduodenitis (Gastrointestinal disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 1
Ophthalmic herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral artery occlusion (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=59)
Blepharitis (Eye disorders) | 4
Conjunctivitis (Eye disorders) | 5
Dry eye (Eye disorders) | 6
Growth of eyelashes (Eye disorders) | 5
Vision blurred (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 35
Gingivitis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 8
Fatigue (General disorders) | 19
Influenza like illness (General disorders) | 9
Pain (General disorders) | 5
Pyrexia (General disorders) | 7
Eye infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 4
Paronychia (Infections and infestations) | 7
Tooth infection (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 6
Blood bilirubin increased (Investigations) | 3
Carcinoembryonic antigen increased (Investigations) | 3
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 5
Pelvic pain (Reproductive system and breast disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 16
Hirsutism (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 55
Dyspepsia (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.